CLINICAL TRIAL: NCT04692129
Title: Short-term Effects of Prone Positioning on Tissue Oxygen Saturation, Measured by Near-infrared Spectroscopy, in COVID-19 Patients With Acute Respiratory Distress Syndrome
Brief Title: Prone Positioning Short-term Effects on Tissue Oxygen Saturation in Critical COVID-19 Patients
Acronym: PRONECOVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Institut de Ciències Fotòniques (ICFO) (Unknown); Centre de Recerca Matemàtica (Unknown); Institute of Physics University of Campinas (Unknown)
Responsible Party: Principal Investigator, Jaume Mesquida, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: 2020/591
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Covid19; ARDS, Human
Keywords: COVID-19; Tissue oxygenation; ARDS; Prone position
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to monitor short-term changes in tissue oxygen saturation and local blood flow as results of changing from supine to prone position in ARDS COVID-19 patients

DETAILED DESCRIPTION:
After obtaining consent to participate in the study, the subjects included in the study will undergo a baseline 15-minute measurement of tissue oxygen saturation (StO2) measured non-invasively on the forearm by means of near-infrared spectroscopy (NIRS). Once a baseline stable StO2 value is obtained, a provocative test, consisting of a transient vascular occlusion, will be performed. The test will allow the obtention of a local metabolic rate, and a StO2 recovery rate after the ischemic stimulus.

Tissue oxygenation measurements will be performed in supine position, immediately before changing to prone positioning, and repeated after 20 minutes of stabilization, once in prone position.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients admitted in the ICU receiving invasive mechanical ventilation and requiring prone positioning for severe hypoxemia management, as decided by the medical team

Exclusion Criteria:

* Severe peripheral vasculopathy
* Raynaud's syndrome
* Skin lesions/trauma in upper limbs interfering the placement of the NIRS probe and/or the occlusion tourniquet
* Deep venous thrombosis in the upper limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients with severe hypoxemia, under mechanical ventilation, and requiring prone positioning as a rescue therapy for hypoxemia management
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in tissue oxygenation (StO2) | 20 minutes
  Tissue oxygenation is measured as percent of oxyhemoglobin over total hemoglobin content in the sensed area (skeletal muscle)
Change in local hemoglobin content (THC) | 20 minutes
  THC is measured as microMols

SECONDARY OUTCOMES:
Compare changes in tissue oxygenation (StO2) and arterial oxygenation (SaO2) | 20 minutes
  Arterial oxygenation (SaO2) is obtained from blood gas analysis, from an arterial blood sample, while StO2 is derived from the sensed tissue, by means of NIRS/DCS technology

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Mesquida, Principal Investigator — Parc Taulí Hospital Universitari
Locations (6):
- Hospital de Clñinicas da UNICAMP, Campinas, São Paulo, Brazil
- Hospital General de México, México, Mexico
- Spain (4):
  - Parc Taulí Hospital Universitari, Sabadell, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Parc Salut Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona